CLINICAL TRIAL: NCT02726555
Title: Comparison Between Combined Therapy With Red Yeast Rice and Low-dose Statin and Standardized Statin: a Single-center, Non-inferiority, Randomized Clinical Trial
Brief Title: The Efficacy and Safety of Combined Therapy With Red Yeast Rice and Low-dose Statin：Comparing With Standardized Statin
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kangting Ji, MD, Professor of Medicine, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: wzfeyxzk
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Dyslipidemia; Atherosclerosis
Keywords: Red yeast rice; Atorvastatin; Mild cardiovascular disease
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis | interventions — red yeast rice; Atorvastatin; xuezhikang

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red yeast rice and atorvastatin (Experimental): Participants will receive 4 identically appearing capsules twice daily for 24 weeks: 2 300mg of red yeast rice and 2 10mg of atorvastatin.
  Interventions: Drug: Red yeast rice and atorvastatin
- Atorvastatin alone (Active Comparator): Participants will receive 4 identically appearing capsules twice daily for 24 weeks: 2 placebo and 2 10mg of atorvastatin.
  Interventions: Drug: Atorvastatin alone

INTERVENTIONS:
Drug: Red yeast rice and atorvastatin — Participants will receive 2 capsules of 300mg red yeast rice and 2 capsules of 10mg atorvastatin for 24 weeks.
  Other Names: Xuezhikang; Lipitor
  Arms: Red yeast rice and atorvastatin
Drug: Atorvastatin alone — Participants will receive 2 capsules of placebo and 2 capsules of 10mg atorvastatin for 24 weeks.
  Other Names: Lipitor
  Arms: Atorvastatin alone

SUMMARY:
Double-dose statin regimen achieves merely 6% of decrease in low-density lipoprotein cholesterol (LDL-C) levels, whereas the risk of side effects increased largely. The investigators' previous pilot study (NCT01686451) has suggested that red yeast rice was of similar lipid-lowering efficacy while was associated with less fatigue than statins. The purpose of this study is to evaluate the efficacy and safety of combined therapy with red yeast rice and low-dose atorvastatin in persons with mild atherosclerotic cardiovascular disease and who qualified for statin therapy according to national guidelines.

DETAILED DESCRIPTION:
Both Red Yeast Rice and Statins are cholesterol-lowering medications are often prescribed for secondary prevention of cardiovascular disease (CVD). The investigators' previous pilot study (NCT01686451) has suggested that red yeast rice was of similar lipid-lowering efficacy while was associated with less fatigue than statins. The aim of this study is to compare the efficacy and safety of combined therapy with red yeast rice at 1.2 g/day and atorvastatin at 10 mg/day with atorvastatin at 20 mg/day in persons with mild atherosclerotic cardiovascular disease and who qualified for statin therapy according to national guidelines.

This study will enroll individuals with established mild atherosclerotic cardiovascular disease and who do not currently take lipid-lowering medications. Participants will be randomly assigned to receive combined therapy with red yeast rice at 1.2 g/day and atorvastatin at 10 mg/day or atorvastatin at 20 mg/day for 24 weeks. Study visits will occur at screening, baseline, week 4, week 8, week 16, and week 24. Blood will be collected for laboratory testing, and standardized questionnaires will assess noncardiovascular endpoints. Pill count will be used to assess adherence of treatment. Medication side effects will be monitored and tests of alanine aminotransferase (ALT), aspartate aminotransaminase (AST) and creatine phosphate kinase (CPK) will be performed. Medication efficacy will be assessed and test of low-density lipoprotein cholesterol (LDL-C) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with established mild atherosclerotic cardiovascular disease, defined as coronary and/or carotid and/or peripheral artery lesions <40% lumen diameter stenosis, diagnosed by coronary angiography and carotid and/or peripheral artery ultrasound respectively, together with LDL cholesterol level > 70 mg/dL (1.80 mmol/L).
2. Female patients must be postmenopausal as defined by no menstruation for at least 12 months, or surgically sterilized for at least three months prior to beginning the study, or have a negative pregnancy test and agree to avoid pregnancy during the study and one month after the end of the study by using two reliable methods of contraception.
3. Patients must have been informed of all aspects of the study and signed an informed consent form before any study-related activities.
4. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Patients who have met all the above inclusion criteria will be screened for the following exclusion criteria.

1. Patients who have been taken lipid-lowering medications including statins or red yeast rice products during the 4 weeks prior to the screening visit.
2. Documented history of myocardial infarction (MI), unstable angina leading to hospitalization, uncontrolled cardiac arrhythmia, percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG), carotid surgery or stenting, cerebrovascular accident, transient ischemic attack, endovascular procedure or surgical intervention for peripheral vascular disease.
3. Planned to undergo scheduled PCI, CABG, carotid or peripheral revascularization during the study.
4. History of New York Heart Association Class III or IV heart failure within the past 12 months.
5. Known history of hemorrhagic stroke.
6. Patients with uncontrolled hypertension at the screening visit. Patients on stable antihypertensive medication may be enrolled provided that the medications and dosage remain stable throughout the study.
7. Cardiovascular surgery or major operations within 6 months prior to screening visit.
8. Patients who are taking anticoagulants except aspirin at < 325 mg/day.
9. Patients with liver dysfunction as indicated by a serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) level of > 1.5-times of upper limit of normal (ULN) range, or clinical symptoms.
10. Patients with elevated creatine phosphokinase level (above Upper Limit of Normal range).
11. Patients with renal dysfunction as indicated by a serum creatinine level above ULN range, or clinical symptoms.
12. Patients with gastric or peptic ulcer within 3 months prior to screening visit.
13. Patients with medical history of hypothyroidism, pancreatitis, cholestasis, nephrotic syndrome, gall bladder disease, or primary biliary cirrhosis. Patients on thyroid replacement therapy at stable doses may be enrolled if clinically euthyroid.
14. Patients with clinically relevant illness within 4 weeks prior to screening visit that may interfere with the conduct of this study.
15. Patients with a history of alcohol or narcotic substance abuse within two years prior to screening visit.
16. Patients with hypersensitivity to lipid-lowering agents.
17. Patients who have taken another investigational drug within 4 weeks prior to screening visit.
18. Patients with uncontrolled metabolic or endocrine disease knowing to influence lipid values.
19. Patients who are known to be HIV positive.
20. Patients who have a history or presence of active malignancy (other than non-melanoma skin cancer) or clinically significant psychiatric, neurological, respiratory, hematological, or other conditions that in the opinion of investigators might interfere with or contraindicate participation of the patients in this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean percentage change from baseline at week 24 (or the last assessment) on serum low-density lipoprotein cholesterol (LDL-C) level | Measured at screening, baseline, week 4, week 8, week 16, and week 24

SECONDARY OUTCOMES:
Mean percentage change from baseline at week 24 (or the last assessment on serum total cholesterol (TC) level | Measured at screening, baseline, week 4, week 8, week 16, and week 24
Mean percentage change from baseline at week 24 (or the last assessment) on serum high-density lipoprotein cholesterol (HDL-C) level | Measured at screening, baseline, week 4, week 8, week 16, and week 24
Mean percentage change from baseline at week 24 (or the last assessment) on serum triglyceride (TG) level | Measured at screening, baseline, week 4, week 8, week 16, and week 24
Mean percentage change from baseline at week 24 (or the last assessment) on serum non-HDL cholesterol level | Measured at screening, baseline, week 4, week 8, week 16, and week 24
Percentage of Participants Who Experienced Statin-associated muscle symptoms (SAMs) | Measured at week 4, week 8, week 16, and week 24
  SAMs included all muscle-related complaints (e.g. pain, weakness, or cramps). Reported events are muscle-related complaints confirmed by an independent Clinical Events Committee (CEC) according to the nature of the muscle symptoms, the elevation in creatine kinase (CK) levels and their temporal association with statin initiation, discontinuation, and re-challenge.

OTHER OUTCOMES:
Mean percentage change from baseline at week 24 (or the last assessment) on serum fasting blood glucose level | Measured at baseline, week 4, week 8, week 16, and week 24
Mean percentage change from baseline at week 24 (or the last assessment) on serum glycosylated hemoglobin level | Measured at baseline, week 4, week 8, week 16, and week 24
Mean percentage change from baseline at week 24 (or the last assessment) on Physical Activity Level | Measured at baseline, week 4, week 8, week 16, and week 24
  Physical activity level will be estimated by short version of international physical activity questionnaire (IPAQ).
Mean percentage change from baseline at week 24 (or the last assessment) on fatigue scores | Measured at baseline, week 4, week 8, week 16, and week 24
  Fatigue score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Mean percentage change from baseline at week 24 (or the last assessment) on Memory problems score | Measured at baseline, week 4, week 8, week 16, and week 24
  Memory problems score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Mean percentage change from baseline at week 24 (or the last assessment) on Attention/concentration problems score | Measured at baseline, week 4, week 8, week 16, and week 24
  Attention/concentration problems score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Mean percentage change from baseline at week 24 (or the last assessment) on Calculation problems score | Measured at baseline, week 4, week 8, week 16, and week 24
  Calculation problems score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Mean percentage change from baseline at week 24 (or the last assessment) on Depression/hopelessness score | Measured at baseline, week 4, week 8, week 16, and week 24
  Depression/hopelessness score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Mean percentage change from baseline at week 24 (or the last assessment) on Anxiety score | Measured at baseline, week 4, week 8, week 16, and week 24
  Anxiety included restless, impatience, irritability, nervous, anxious. Anxiety score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Mean percentage change from baseline at week 24 (or the last assessment) on Sleep problems score | Measured at baseline, week 4, week 8, week 16, and week 24
  Sleep problems score is self-rated, ranging from 0-10. For the severity scale, 0=not present, 10=most severe.
Safety will be assessed by the incidence of adverse events (AEs), discontinuation due to the AEs, clinically relevant changes on laboratory test results, vital signs, physical examinations, and 12-lead electrocardiograms (ECG). | Screening, Baseline, Week 4, Week 8, week 16, and week 24
  ECG and Physical exam only at Screening and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Kangting Ji, MD, Principal Investigator — The Second Hispital of Wenzhou Medical University
Locations (1):
- The Second Hispital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided